CLINICAL TRIAL: NCT04813640
Title: A Prospective, Randomised, Dispensing Clinical Trial to Compare the Visual Performance, Wearability and Ocular Response of Myopia Control, Novel Myopia Control and Single Vision Spectacle Lenses
Brief Title: Eye Length Signal With Myopia Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brien Holden Vision Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCRTC2020-02
Record Dates: First submitted 2021-02-04; First posted 2021-03-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Vision Spectacles (Placebo Comparator): Commercially available conventional single vision spectacles
  Interventions: Device: Spectacles
- Commercially available myopia control spectacles (Active Comparator): Commercially available myopia control spectacles
  Interventions: Device: Spectacles
- Novel Myopia control spectacles - Prototype I (Experimental): Experimental myopia control spectacles
  Interventions: Device: Spectacles
- Novel Myopia control spectacles - Prototype II (Experimental): Experimental myopia control spectacles
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Spectacles — Novel spectacles for myopia control

SUMMARY:
Myopia, considered as a global epidemic, is rapidly rising in prevalence especially in east Asian countries. Younger ages are associated with greater annual progression and thus early onset myopia is likely to result in higher levels of final net myopia.[1] Myopia, especially high myopia (more than -6.00D) is associated vision threatening complications such as cataract, glaucoma, choroidal thinning, vitreous liquefaction, myopic maculopathy, retinal detachment etc. Furthermore, myopia can affect the quality of life of an individual through restriction of employment in certain fields such as aviation. Myopia also imposes economic burden through the recurring cost of vision correction such as spectacles, contact lenses and specialist consultation fee. It is therefore important to develop novel optical and pharmaceutical strategies that can control or slow the progression of myopia.

DETAILED DESCRIPTION:
To date, the strategies used to control or slow the progression of myopia are optical and pharmaceutical methods. Among spectacles, bifocal spectacles with and without prism, progressive addition lenses, spectacles altering peripheral hyperopic defocus, spectacles imposing myopic defocus both centrally and peripherally and spectacles with multiple defocus segments that imposes myopic defocus in front, midperiphery and periphery of the retina (defocus incorporating multiple segments or DIMS) are used to reduce the progression[2-6]. Of these, spectacles designed to alter peripheral defocus demonstrated a small treatment effect in reducing myopia progression[6, 7]. Bifocal and progressive addition spectacles demonstrated variable treatment effect in reducing progression of myopia. Among contact lenses, multifocal contact lenses altering peripheral defocus, extended depth of focus contact lenses altering higher order aberrations in order to degrade the retinal image behind the retina have shown promising results in slowing myopia progression along with orthokeratology treatment[8-12]. Among these, orthokeratology and multifocal soft contact lenses (centre distance multifocal contact lenses) showed promising results in slowing myopia progression[9, 12].

Pharmaceutical interventions include Atropine, Pirenzepine, 7-Methylxanthine and Timolol[13].Atropine is the most widely used, with higher concentrations more effective. Atropine 1% concentration demonstrated 60 to 80% reduction in progression of myopia. However, ocular side effects such as blurred vision, photophobia etc associated with atropine makes it a less appealing option. Among the various treatment approaches, spectacles pose the least or minimal side effects compared to contact lenses, orthokeratology or pharmaceutical strategies. Therefore, this study aims to determine the effect of novel myopia control prototype spectacle design on wearability and physiological ocular response among myopic children aged 7 to 14 years.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 7 to 14 completed years (7 and 14 years inclusive), irrespective of gender.
* have cycloplegic autorefraction spherical component -0.50 D to - 4.50D, cylinder no more than -1.50D
* be accompanied by parents/guardians who can read and comprehend Vietnamese and give informed consent as demonstrated by signing a record of informed consent.
* be willing to comply with the wearing and clinical trial visit schedule as directed by the Investigator.
* have ocular health findings considered to be "normal".
* be correctable to at least 6/9.5 (20/30) or better in each eye with spectacles.
* be willing to wear the spectacles provided by the investigators for all waking hours;

Exclusion Criteria:

* A known allergy to, or a history of intolerance to tropicamide or topical anaesthetics;
* Strabismus and/or amblyopia;
* Had previous eye surgery (including strabismus surgery);
* Any ocular, systemic or other condition or disease with possible associations with myopia or affecting refractive development e.g. Marfan syndrome, retinopathy of prematurity, diabetes;
* Had any ocular injury or condition (including keratoconus and herpes keratitis) of the cornea, conjunctiva or eyelids;
* Worn bifocals or progressive addition spectacles;
* Worn orthokeratology or bifocal contact lenses;
* Current orthoptic treatment or vision training;
* Any anatomical, skin or other condition that would impact on the wearing of spectacles;
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Concurrently enrolled in another clinical trial.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in axial length | one monthly interval for up to 6 months
  Change in axial length measured using Lenstar

SECONDARY OUTCOMES:
Vision and Choroidal Physiology | One monthly interval for up to 6 months
  Vision and Choroidal Physiology determined using standard vision charts and Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Minh Huy Tran, M.D., Msc., Principal Investigator — Hai Yen Eye Care
Locations (1):
- Hai Yen Eye Care Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No